CLINICAL TRIAL: NCT00705458
Title: A Randomized Trial Comparing Multi-Detector Coronary CT Angiography and Stress Myocardial Perfusion Imaging as the Initial Test for the Diagnosis of Coronary Artery Disease in Intermediate Risk Patients Admitted for Chest Pain
Brief Title: Study Comparing CT Scan and Stress Test in Diagnosing Coronary Artery Disease in Patients Hospitalized for Chest Pain
Acronym: PROSPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: American Heart Association (Other); Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Jeffrey Levsky, Associate Director of Research, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MMC-07-07-197
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Unstable Angina; Acute Coronary Syndrome
Keywords: stress myocardial perfusion imaging; coronary computed tomography angiography
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Angina, Unstable; Acute Coronary Syndrome | interventions — Exercise Test; Technetium Tc 99m Sestamibi; Thallium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CTA (Experimental): Initial EKG-gated computed tomography angiography of the coronary arteries
  Interventions: Procedure: Coronary Computed Tomography Angiography
- MPI (Active Comparator): Initial nuclear stress myocardial perfusion imaging
  Interventions: Procedure: Stress Nuclear Myocardial Perfusion Imaging

INTERVENTIONS:
Procedure: Coronary Computed Tomography Angiography — 64-detector, retrospectively EKG-gated, computed tomography angiography of the coronary arteries during heart rate control (intravenous metoprolol, when necessary)
  Other Names: CCTA; Coronary CT; Coronary CTA; Coronary Artery CT; Coronary Artery CTA; Coronary CT Angiography; CTA of the Coronary Arteries
  Arms: CTA
Procedure: Stress Nuclear Myocardial Perfusion Imaging — Usually dual-isotope perfusion imaging at rest (201-Thallium) and at stress (99m-Technetium-MIBI). Some patients will have a 2-day MIBI protocol. Gated SPECT and attenuation-correction images will be obtained. Treadmill stress will be performed. If a patient is unable to exercise, adenosine or dobutamine will be given.
  Other Names: stress test; nuclear stress test; dual-isotope stress test; sestamibi; thallium; myocardial perfusion imaging; nuclear perfusion imaging; gated SPECT; nuclear cardiology
  Arms: MPI

SUMMARY:
The purpose of this study is to determine whether coronary artery CT scanning or nuclear stress testing is better at diagnosing chest pain patients with coronary artery disease to select appropriate candidates for coronary catheterization and re-vascularization.

ELIGIBILITY:
Inclusion Criteria:

* patient admitted for chest pain or pressure
* patient at intermediate short term risk of MI or death (AHA/ACC guidelines)

Exclusion Criteria:

* prior diagnosis of coronary artery disease
* evidence of ongoing myocardial infarction (and other high risk criteria per AHA/ACC guidelines)
* contraindications to EKG-gated CT scanning with iodinated intravenous contrast under beta-blockade
* pregnancy
* presence of an implanted pacemaker or defibrillator
* stress myocardial perfusion imaging, coronary CTA or coronary catheterization within the last 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2008-07; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Coronary catheterization that does not lead to re-vascularization | 1 year

SECONDARY OUTCOMES:
Length of Hospital Stay (time to discharge) | usually from hours to a few days (average about one day)
Non-fatal myocardial infarction | 1 year
Death (all cause) | 1 year
Post-test renal dysfunction | usually within a few days

CONTACTS AND LOCATIONS:
Overall Officials: Linda B Haramati, MD, MS, Study Director — Montefiore Medical Center/Albert Einstein College of Medicine; Jeffrey M Levsky, MD, PhD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Moses Division, Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Background] Levsky JM, Travin MI, Spevack DM, Menegus MA, Huang PW, Goldberg Y, Clark ET, Banoth P, Freeman KD, Tobin JN, Haramati LB. Rationale and design of a randomized controlled trial comparing stress myocardial perfusion imaging with coronary CT angiography as the initial imaging study for intermediate-risk patients admitted with chest pain. J Cardiovasc Comput Tomogr. 2009 Jul-Aug;3(4):264-71. doi: 10.1016/j.jcct.2009.05.006. Epub 2009 May 21. PMID 19577217
- [Result] Levsky JM, Spevack DM, Travin MI, Menegus MA, Huang PW, Clark ET, Kim CW, Hirschhorn E, Freeman KD, Tobin JN, Haramati LB. Coronary Computed Tomography Angiography Versus Radionuclide Myocardial Perfusion Imaging in Patients With Chest Pain Admitted to Telemetry: A Randomized Trial. Ann Intern Med. 2015 Aug 4;163(3):174-83. doi: 10.7326/M14-2948. PMID 26052677